CLINICAL TRIAL: NCT00780130
Title: The Relationship of Core Stability to Core Proprioception
Brief Title: SPARQ and Core Proprioception
Status: Completed | Type: Observational
Sponsor: Logan College of Chiropractic (Other)
Responsible Party: Dr. Dennis Enix, Logan College of Chiropractic
Other Study IDs: RD1028080161
Record Dates: First submitted 2008-10-22; First posted 2008-10-27 (Estimated); Last update posted 2008-10-28 (Estimated); Status verified 2008-10

CONDITIONS: Proprioception; Core Strength

STUDY DESIGN:
Observational Model: Case-Only
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1: male & female college students ages 20 to 50, asymptomatic normals
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — male & female college students ages 20 to 50, asymptomatic normals

SUMMARY:
The purpose of this investigation is to determine the relationship of core stability to core proprioception

DETAILED DESCRIPTION:
As no previous research has been reported correlating the SPARQtm method of athletic performance with the McGill Side Bridge test and core joint position error, this study is designed as a pilot. The subject's core stability will be measured with the SPARQtm method of athletic performance and the McGill Side Bridge test for core stability. Core proprioception will be determined using the standard test for proprioception, Joint Position Error (JPE) testing, with the Skill Technologies motion capture device. All participants will receive the SPARQtm method of athletic performance testing, the McGill Side Bridge test for core stability and the core joint position error tests twice, one week apart.

ELIGIBILITY:
Inclusion Criteria:

* college student, staff, or faculty members;
* History of thoracic / lumbar injuries for inclusion into the injured group.
* No history of thoracic / lumbar injuries for inclusion into the normal group.
* Ages 20 to 50
* History of previous athletic performance.

Exclusion Criteria:

* Previous lower extremity injury, surgery, visual or vestibular condition affecting balance
* Current acute illness that have an adverse effect on balance or core strength
* Local infection, injury or other malignancy
* Any unstable joints of the lower extremity or spine
* Any Spinal manipulation within 48 hours
* Prescription medication or supplement that affects blood pressure
* Pregnancy
* Diagnosis of severe hypertension (200-161/120-100 mmHg)
* Incapable of exercise for 15 minutes without hortness of breath
* Heart failure, kidney diseases and mental disorders

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: asymptomatic normals
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2008-05; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Mcgill sidebridge test proprioception testing SPARQ testing | Two testing sessions one week apart.

CONTACTS AND LOCATIONS:
Locations (1):
- Logan College of Chiropractic, Chesterfield, Missouri, United States